CLINICAL TRIAL: NCT01347827
Title: Comparison of Cerebral Tissue Oxygen Desaturation in Patients Undergoing On-pump or Off-pump Coronary Artery Bypass Grafting
Brief Title: Tissue Oxygenation During Heart Surgery
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: TO-CABG
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Coronary artery bypass surgery; Oximetry; Brain metabolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- on pump: Coronary artery bypass grafting (CABG)with with cardiopulmonary bypass
  Interventions: Device: measurements of brain tissue oxygenation
- off pump: off-pump CABG surgery
  Interventions: Device: measurements of brain tissue oxygenation

INTERVENTIONS:
Device: measurements of brain tissue oxygenation — different monitors((the Hutchinson InSpectra™ StO2 Tissue Oxygenation Monitor) and in cerebral (ForeSight® Cerebral Oximeter and the Somanetics INVOS® Cerebral Oximeter ) and renal tissue (the Somanetics INVOS® Cerebral Oximeter)of brain tissue oxygenation with each other, and assess the correlation between brain tissue oxygenation and oxygenation measurements in renal and muscular tissue, as well as with conventional hemodynamic and metabolic variables, such as central venous oxygen saturation
  Groups: on pump
Device: measurements of brain tissue oxygenation — different monitors((the Hutchinson InSpectra™ StO2 Tissue Oxygenation Monitor) and in cerebral (ForeSight® Cerebral Oximeter and the Somanetics INVOS® Cerebral Oximeter ) and renal tissue (the Somanetics INVOS® Cerebral Oximeter) of brain tissue oxygenation with each other, and assess the correlation between brain tissue oxygenation and oxygenation measurements in renal and muscular tissue, as well as with conventional hemodynamic and metabolic variables, such as central venous oxygen saturation
  Groups: off pump

SUMMARY:
The goal of this study is to determine if off-pump CABG surgery is associated with better cerebral tissue oxygenation when compared with on-pump CABG. In addition, the investigators would like to compare the results of two different monitors of brain tissue oxygenation with each other, and assess the correlation between brain tissue oxygenation and oxygenation measurements in renal and muscular tissue, as well as with conventional hemodynamic and metabolic variables, such as central venous oxygen saturation (ScvO2). Finally, the investigators aim to determine if duration and extent of cerebral oxygen desaturation predict outcome variables such as postoperative cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed patient consent
* Coronary artery disease suitable for both on-pump and off-pump CABG surgery.

Exclusion Criteria:

* History of head trauma or stroke causing significant active neurologic disease
* History of neurosurgery
* Severe or symptomatic carotid artery disease
* Requirement for valve surgery in addition to CABG
* Pre-existing acute or chronic renal dysfunction
* Urgent or emergency surgery
* Difficulty with cognitive testing: impaired hearing or eyesight, poor Dutch language comprehension, disability impairing the usage of the hand or arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 consecutive adult patients scheduled for elective CABG surgery will be randomized to have the surgery performed either on-pump (n=30) or off-pump CABG (n=30).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
incidence of significant brain tissue oxygen desaturation, defined as AUC40 > 600 %.sec (a function of both duration (in seconds) and severity (saturation < 40%) of desaturation). | 3 months

SECONDARY OUTCOMES:
Oxygenation measurements: Peripheral muscle StO2, cerebral and renal StO2, ScvO2, SaO2, arteriovenous oxygen difference, pO2 Acid-base status: pH, pCO2, HCO3-, ABE, lactate | 3 months
  * To determine if oxygenation measurements obtained in peripheral (thenar) muscle, renal tissue and in cerebral tissue correlate with each other
  * To determine if oxygenation measurements obtained in peripheral (thenar) muscle, renal tissue and in cerebral tissue correlate with conventional hemodynamic and metabolic variables such as central venous oxygen saturation (ScvO2).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W.L. Scheeren, Prof.dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] de Keijzer IN, Poterman M, Absalom AR, Vos JJ, Mariani MA, Scheeren TWL. Comparison of renal region, cerebral and peripheral oxygenation for predicting postoperative renal impairment after CABG. J Clin Monit Comput. 2022 Jun;36(3):735-743. doi: 10.1007/s10877-021-00701-4. Epub 2021 Apr 20. PMID 33876337